CLINICAL TRIAL: NCT02932332
Title: High-Flow Oxygen for Dyspnea in Hospitalized Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-0282; NCI-2017-00186 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Cancer
Keywords: shortness of breath; oxygen; breathing therapies
MeSH Terms: conditions — Neoplasms; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- High-flow oxygen: Initial Therapy (Active Comparator): 4-Period crossover therapy where initial 10 minute breathing treatment with High-flow oxygen (HFOx) is followed by 3 different breathing therapies of Low-flow oxygen (LFOx), High-flow air (HFAir), and Low-flow air (LFAir) with 10 minute washout period before subsequent treatments for a total 80 minute study period accompanied by shortness of breath questionnaires.
  Interventions: Other: High-flow Oxygen; Other: Low-flow Oxygen; Other: High-flow Air; Other: Low-flow Air
- Low-flow oxygen: Initial Therapy (Active Comparator): 4-Period crossover therapy where initial 10 minute breathing treatment with Low-flow oxygen (LFOx) is followed by 3 different breathing therapies of HFOx, HFAir, and LFAir with 10 minute washout period before subsequent treatments for a total 80 minute study period accompanied by shortness of breath questionnaires.
  Interventions: Other: High-flow Oxygen; Other: Low-flow Oxygen; Other: High-flow Air; Other: Low-flow Air
- High-flow air: Initial Therapy (Sham Comparator): 4-Period crossover therapy where initial 10 minute breathing treatment with High-flow oxygen (LFOx) is followed by 3 different breathing therapies of HFOx, LFOx, and LFAir with 10 minute washout period before subsequent treatments for a total 80 minute study period accompanied by shortness of breath questionnaires.
  Interventions: Other: High-flow Oxygen; Other: Low-flow Oxygen; Other: High-flow Air; Other: Low-flow Air
- Low-flow air: Initial Therapy (Sham Comparator): 4-Period crossover therapy where initial 10 minute breathing treatment with Low-flow air (LFAir) is followed by 3 different breathing therapies of HFOx, LFOx, and HFAir with 10 minute washout period before subsequent treatments for a total 80 minute study period accompanied by shortness of breath questionnaires.
  Interventions: Other: High-flow Oxygen; Other: Low-flow Oxygen; Other: High-flow Air; Other: Low-flow Air

INTERVENTIONS:
Other: High-flow Oxygen — Optiflow Respiratory Humidifier used to deliver HFOx. Oxygen flow will be maximized (set between 20 and 60 L/min), if tolerated, to minimize dyspnea. FiO2 will be set at 100%.
  Other Names: HFOx
Other: Low-flow Oxygen — Low-flow Oxygen will be delivered by Optiflow in an identical manner to high flow, except provided at 2 L/min using a nasal cannula identical to that used for high-flow devices.
  Other Names: LFOx
Other: High-flow Air — Two level air flow (high and low) will be delivered by Optiflow in an identical manner to oxygen air flows, except that researchers will use pressurized air instead of oxygen. LFOx and LFAir will be provided at 2 L/min using a nasal cannula identical to that used for high-flow devices.
  Other Names: HFAir
Other: Low-flow Air — Two level air flow (high and low) will be delivered by Optiflow in an identical manner to oxygen air flows, except that researchers will use pressurized air instead of oxygen. LFOx and LFAir will be provided at 2 L/min using a nasal cannula identical to that used for high-flow devices.
  Other Names: LFAir

SUMMARY:
The goal of this clinical research study is to compare high-flow oxygen, low-flow oxygen, high-flow air, and low-flow air in helping to decrease shortness of breath in cancer patients. Researchers also want to learn if these therapies can help to improve lung function and quality of life.

DETAILED DESCRIPTION:
Study Groups and Procedures:

If you agree to take part in this study, you will receive 4 different breathing therapies:

* High-flow oxygen
* Low-flow oxygen
* High-flow air and
* Low-flow air

The order in which they will be given to you will be randomly assigned (as in a roll of dice). You will have an equal chance of being assigned to each group. Neither you nor the study staff will know which therapy order you are assigned to. However, if needed for your safety, the study staff will be able to find out what you are receiving.

All 4 breathing therapies should take about 80 minutes total to complete (10 minutes for each treatment with a 10 minute break between each treatment). You will receive the air or oxygen through small tubes placed in your nose. The respiratory therapist will be there to adjust the therapy to your comfort level.

At the end of each breathing therapy, you will be asked about your shortness of breath and if you have any improvement. You will also be asked if you could tell whether you received oxygen or air after each therapy.

After finishing the 4 breathing therapies, you will complete 2 questionnaires about which breathing therapy you liked and your thoughts about taking part in the study. These should take about 10 minutes total to complete.

Length of Study:

You will be taken off study if you no longer wish to take part, or if you need drugs to help with shortness of breath during the study. Your participation in the study will be over after you complete the questionnaires.

This is an investigational study. Comparing high-flow air, low-flow air, high-flow oxygen, and low-flow oxygen to treat shortness of breath is considered investigational.

Up to 36 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer
2. Patients seen by palliative care, thoracic oncology, pulmonary medicine, or emergency care at MD Anderson Cancer Center
3. Dyspnea Numeric Rating Scale at rest >/=3 of 10 (average over last 24 hour)
4. Non-hypoxemic (i.e. oxygen saturation >90% on ambient air)
5. Able to communicate in English or Spanish
6. Age >/= 18 years
7. Able to tolerate high-flow oxygen/air

Exclusion Criteria:

1. Memorial Delirium Rating Scale >13
2. Hemodynamic instability
3. Respiratory failure requiring mechanical ventilation or non-invasive ventilation
4. Frequent use of rescue opioids >8x/day or rescue bronchodilators >8x/day over last 24 hours
5. Currently requiring high flow oxygen for oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Hernandez F, Urbauer D, Thomas S, Lu Z, Elsayem A, Bruera E. High-Flow Oxygen and High-Flow Air for Dyspnea in Hospitalized Patients with Cancer: A Pilot Crossover Randomized Clinical Trial. Oncologist. 2021 May;26(5):e883-e892. doi: 10.1002/onco.13622. Epub 2020 Dec 15. PMID 33289276
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from MD Anderson Cancer Center with active cancer diagnosis , having age >=18, an average dyspnea numeric rating scale of ≥4/10 over the past 24 hours, oxygen saturation >90% on ambient air and able to tolerate high flow nasal canula.
Pre-assignment Details: 19 patients were randomized for this study. 7 patients were not randomized for various reasons (discharged too early=3, changed mind=2 and others =2)
Groups:
- Group 1 High Flow Air (HFAir-LFAir-HFOx-LFOx); Group 2 High Flow Oxygen (HFOx-HFAir-LFOx-LFAir); Group 3 Low Flow Air (LFAir-LFOx-HFAir-HFOx); Group 4 Low Flow Oxygen (LFOx-HFOx-LFAir-HFAir): High Flow Oxygen and High Flow Air was delivered between 20 and 60 L/min. Low Flow Oxygen and Low Flow Air was delivered at 2L/min
Period: Overall Study
Arm/Group | Group 1 High Flow Air (HFAir-LFAir-HFOx-LFOx) | Group 2 High Flow Oxygen (HFOx-HFAir-LFOx-LFAir) | Group 3 Low Flow Air (LFAir-LFOx-HFAir-HFOx) | Group 4 Low Flow Oxygen (LFOx-HFOx-LFAir-HFAir)
Started | 5 | 4 | 5 | 5
Intervention 1 | 4 | 4 | 5 | 4
Intervention 2 | 4 | 3 | 4 | 4
Intervention 3 | 3 | 2 | 4 | 3
Intervention 4 | 3 | 1 | 4 | 3
Completed | 3 | 1 | 4 | 3
Not Completed | 2 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Chest pain | 0 | 0 | 0 | 1
Not completed — Not Dyspneic cough | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: It included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 High Flow Air (HFAir-LFAir-HFOx-LFOx) | Group 2 High Flow Oxygen (HFOx-HFAir-LFOx-LFAir) | Group 3 Low Flow Air (LFAir-LFOx-HFAir-HFOx) | Group 4 Low Flow Oxygen (LFOx-HFOx-LFAir-HFAir) | Total
Number analyzed (Participants) | 5 | 4 | 5 | 5 | 19
Age, Continuous [Mean (Full Range); unit: years] | 55 [35 to 68] | 48 [29 to 62] | 50 [36 to 59] | 51 [34 to 70] | 51 [29 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 3 | 11
  Male | 3 | 1 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 4 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 4 | 3 | 3 | 5 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 5 | 5 | 19
Cancer Stage [Count of Participants; unit: Participants] — Cancer is typically labeled in stages from I to IV, with IV being the most serious.
  Participants
    II | 0 | 0 | 0 | 1 | 1
    III | 0 | 0 | 1 | 0 | 1
    IV | 5 | 4 | 4 | 4 | 17
Cancer Type [Count of Participants; unit: Participants]
  Breast | 0 | 0 | 1 | 1 | 2
  Gastrointestinal | 3 | 1 | 1 | 2 | 7
  Genitourinary | 0 | 1 | 1 | 0 | 2
  Gynecological | 0 | 0 | 1 | 0 | 1
  Hematologic | 0 | 1 | 0 | 1 | 2
  Thoracic | 1 | 1 | 1 | 1 | 4
  Other | 1 | 0 | 0 | 0 | 1
Dyspnea for reason of admission [Count of Participants; unit: Participants]
  Yes | 2 | 1 | 4 | 2 | 9
  No | 3 | 3 | 1 | 3 | 10
Supplement Oxygen [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 3 | 2 | 9
  No | 2 | 3 | 2 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Dyspnea Numeric Score Between 0 and 10 Minutes
Description: We assessed dyspnea intensity 'now' using a numeric rating scale from 0 to 10 where 0=none and 10=worst. The minimal clinically important difference was 1 point.
Time Frame: 0 (baseline) minutes and at 10 minutes
Population: Participants who completed the first intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 High Flow Air (HFAir-LFAir-HFOx-LFOx) | Group 2 High Flow Oxygen (HFOx-HFAir-LFOx-LFAir) | Group 3 Low Flow Air (LFAir-LFOx-HFAir-HFOx) | Group 4 Low Flow Oxygen (LFOx-HFOx-LFAir-HFAir)
Number analyzed (Participants) | 4 | 4 | 5 | 4
score on a scale | -1.8 [-3.0 to -0.5] | -1.8 [-2.8 to -0.7] | -0.6 [-1.3 to 0.2] | -0.5 [-1.0 to 0.1]

2. Secondary Outcome: Change in Modified Borg Scale Intensity Between 0 and 10 Minutes
Description: We assessed dyspnea intensity 'now' using a Modified Dyspnea Borg scale. This is a 0-10 point ratio scale with a higher score indicating worse dyspnea.
Time Frame: 0 (baseline) minutes and at 10 minutes
Population: Participants who completed the first intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 High Flow Air (HFAir-LFAir-HFOx-LFOx) | Group 2 High Flow Oxygen (HFOx-HFAir-LFOx-LFAir) | Group 3 Low Flow Air (LFAir-LFOx-HFAir-HFOx) | Group 4 Low Flow Oxygen (LFOx-HFOx-LFAir-HFAir)
Number analyzed (Participants) | 4 | 4 | 5 | 4
score on a scale | -0.7 [-1.6 to 0.2] | -1.8 [-2.8 to -0.7] | -0.1 [-0.4 to 0.2] | -0.5 [-1.2 to 0.2]

3. Secondary Outcome: Change in Modified Borg Scale Unpleasantness Between 0 and 10 Minutes
Description: We assessed dyspnea unpleasantness 'now' using a Modified Dyspnea Borg scale. This is a 0-10 point ratio scale with a higher score indicating worse dyspnea unpleasantness.
Time Frame: 0 (baseline) minutes and at 10 minutes
Population: Participants who completed the first intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 High Flow Air (HFAir-LFAir-HFOx-LFOx) | Group 2 High Flow Oxygen (HFOx-HFAir-LFOx-LFAir) | Group 3 Low Flow Air (LFAir-LFOx-HFAir-HFOx) | Group 4 Low Flow Oxygen (LFOx-HFOx-LFAir-HFAir)
Number analyzed (Participants) | 4 | 4 | 5 | 4
score on a scale | -0.5 [-1.6 to 0.5] | -1.8 [-3.3 to -0.4] | -0.6 [-1.5 to 0.2] | -0.7 [-1.6 to 0.2]

ADVERSE EVENTS:
Time Frame: baseline and 10 minutes of each intervention.
Description: Adverse effects such as dry eyes, dry nose, nasal moisture and anxiety were assessed using a 0-10 numeric rating scale, where 0=none and 10=worst possible. The participants 'at risk' are a total number of participants combined that received specific intervention from each group at different sequences.
Groups:
- High Flow Air: High Flow Air was delivered between 20 and 60 L/min.
- High Flow Oxygen: High Flow Oxygen was delivered between 20 and 60 L/min.
- Low Flow Air: Low Flow Air was delivered at 2L/min.
- Low Flow Oxygen: Low Flow Oxygen was delivered at 2L/min.
Arm/Group | High Flow Air | High Flow Oxygen | Low Flow Air | Low Flow Oxygen
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 7/12 | 6/13 | 4/13 | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Flow Air (N=12) | High Flow Oxygen (N=13) | Low Flow Air (N=13) | Low Flow Oxygen (N=13)
Dry Nose (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 7
Moisture in nose (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 2 | 5
Nasal prong uncomfortable (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3 | 5
Anxiety (Nervous system disorders) | 4 | 3 | 4 | 1
Feeling of suffocation (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 0
Trouble talking (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 2
Dry eyes (Nervous system disorders) | 1 | 2 | 1 | 1
Eye irritation (Nervous system disorders) | 0 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT02932332/Prot_SAP_000.pdf